CLINICAL TRIAL: NCT04601987
Title: Healthy Moms: Prenatal Counseling for Postpartum Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1623168
Record Dates: First submitted 2020-08-18; First posted 2020-10-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related; Breastfeeding; Maternal Care Patterns
Keywords: Pregnant, breastfeeding, smokefree
MeSH Terms: conditions — Breast Feeding | interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling about the Maternal Benefits of Breastfeeding (Active Comparator): Participants will review a slide deck while receiving scripted counseling designed to increase understanding of the maternal health benefits of breastfeeding.
  Interventions: Behavioral: Breastfeeding
- Counseling about the benefits of Smoke-free Homes (Active Comparator): Participants will review a slide deck while receiving scripted counseling designed to increase understanding of the health benefits of smoke free homes.
  Interventions: Behavioral: Smokefree Homes

INTERVENTIONS:
Behavioral: Breastfeeding — Counseling about the maternal health benefits of lactation.
  Arms: Counseling about the Maternal Benefits of Breastfeeding
Behavioral: Smokefree Homes — Counseling about the importance of smoke-free homes.
  Arms: Counseling about the benefits of Smoke-free Homes

SUMMARY:
See https://studypages.com/s/healthy-moms-study-765273

This individual-level randomized trial involves pregnant women followed for at least 6 months after delivery, to compare the effects of providing two "attention-control" counseling interventions designed to increase pregnant women's awareness of either:

1. the maternal health benefits of breastfeeding, or
2. the health benefits of smoke-free homes

DETAILED DESCRIPTION:
The investigators will conduct an individual-level randomized trial involving pregnant women to compare the effects on infant feeding practices of providing pregnant women information about the maternal health benefits of breastfeeding to usual prenatal counseling focused on the infant health benefits of breastfeeding. Participants will be randomly allocated to one of two equal sized groups by research assistants using a web-based random number generator that conceals allocation. Participants will be recruited online via UC Davis' StudyPages website. Screening will occur online at the participant's convenience. When screening criteria have been met, the research coordinator will be notified, and initiate contact with the participant by text and/or phone call to schedule a time to deliver the intervention. Due to social distancing measures that have been put into place as a result of the COVID-19 pandemic, informed consent will be collected digitally using the Qualtrics platform after potential participants complete a secondary screening survey. Consenting participants will use Qualtrics to complete a baseline/enrollment survey and be randomized and then scheduled for a time to receive their allocated counseling intervention using the Zoom platform. Follow-up surveys will be distributed to participants at 1, 3, 6, 9 and 12 months postpartum.

Comparators:

Participants randomized to the "intervention group" will receive information about the maternal health benefits of breastfeeding from a research assistant who also will provide information on resources designed to support prenatal and postpartum health, including breastfeeding support groups. Participants will be presented with a series of images to look at while listening to the scripted counseling, including an image developed in 2002 by the Ad Council designed to convey a link between bottle-feeding and insulin use, as well as images developed specifically for use when counseling women about the maternal benefits of breastfeeding.

The "attention control" group will receive "usual care" from their prenatal care provider that focuses on the infant health benefits of breastfeeding. To control for the potential effects of receiving additional attention from a counselor, pregnant women enrolled in the control arm of this study will receive information from a peer counselor on the health benefits of "smoke- and weed-free homes".

The investigators will thoroughly train all research staff on the critical importance of delivering only the allocated counseling intervention to each study participant. The investigators will monitor intervention delivery by audio-recording staff interactions with study participants, and providing prompt feedback to research staff, if needed.

Intervention Delivery: These scripted counseling interventions were designed to be understood by those with no more than a fifth-grade education and to take less than 5 minutes to deliver. All research staff will be trained by the PI to ensure they understand the importance of maintaining the integrity of study group allocation and delivering only the assigned scripted counseling. After receiving their allocated counseling, participants will be emailed the images and script and encouraged to share this information with the people they anticipate receiving postpartum support from.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women who are carrying a singleton pregnancy between 27-37 weeks gestation
* Born in the United States
* Aged 18-40 years
* Able to read English
* Have reliable access to a telephone that is able to send and receive text messages
* Have reliable access to a smart phone, tablet, computer, or other device with access to the internet

Exclusion Criteria:

* Women carrying multiple gestations
* Diagnosed with HIV or are advised by a clinician not to breastfeed for any other reason
* Have undergone mastectomy or breast reduction surgery
* Unable to speak English, or who do not have a telephone or respond to text messages
* Carrying a surrogate pregnancy or are not planning to parent after giving birth
* Became pregnant through use of assisted reproductive technology such as in vitro fertilization (IVF)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nulliparous women
Enrollment: 451 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Duration of breastfeeding | at 6 months postpartum
  Total number of weeks of breastfeeding

SECONDARY OUTCOMES:
Knowledge of the maternal health benefits of lactation | 1 month postpartum
  Change in participant knowledge before and after receipt of this counseling intervention will be assessed by asking participants to respond (true, false, don't know) whether they believe Breastfeeding will…
  1. lower my risk of breast cancer.
  2. lower my risk of ovarian cancer.
  3. lower my risk of developing diabetes.
  4. increase my risk of a breast infection.
  5. increase my risk of depression [reverse coded]
  6. make it harder to "get my body back" after my baby is born. [reverse coded]
  7. protect my hands from arthritis.
  8. lower my blood pressure and risk of heart disease.
  9. lower my libido/sex drive.
  10. delay my menstrual period after my baby is born.
  11. save my family money."
Smoke-free home policy | 6 months postpartum
  Investigators will compare the proportion of individuals who have a "smoke-free" policy for their homes as assessed by responding with option "d" when presented with the following options "Which of the following statements best describes the rules about smoking inside your home now, even if no one who lives in your home is a smoker? Select ONE answer
  1. Smoking is permitted anywhere inside my home
  2. Smoking is permitted inside my home by an open window
  3. Smoking is allowed in some rooms or at some times
  4. No one is allowed to smoke anywhere inside my home
Smoke-free home policy | 1 month postpartum
  Investigators will compare the proportion of individuals who have a "smoke-free" policy for their homes as assessed by responding with option "d" when presented with the following options "Which of the following statements best describes the rules about smoking inside your home now, even if no one who lives in your home is a smoker? Select ONE answer
  1. Smoking is permitted anywhere inside my home
  2. Smoking is permitted inside my home by an open window
  3. Smoking is allowed in some rooms or at some times
  4. No one is allowed to smoke anywhere inside my home
Duration of any breastfeeding or pumping at 24 months postpartum | 24 months postpartum
  Investigators will compare the duration of any breastfeeding or pumping reported through 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Bimla Schwarz, MD, MS, Principal Investigator — UC Davis Health
Locations (1):
- UC Davis Center for Healthcare Policy and Research, Sacramento, California, United States

REFERENCES:
- [Result] Schwarz EB, Hoyt-Austin A, Fix M, Kair LR, Iwuagwu C, Chen MJ. Prenatal Counseling on the Maternal Health Benefits of Lactation: A Randomized Trial. Breastfeed Med. 2024 Jan;19(1):52-58. doi: 10.1089/bfm.2023.0219. Epub 2024 Jan 8. PMID 38190278
- [Result] Iwuagwu C, Chen MJ, Hoyt-Austin AE, Kair L, Fix M, Schwarz EB. Awareness of the Maternal Health Benefits of Lactation Among U.S. Pregnant Individuals. Womens Health Issues. 2024 May-Jun;34(3):283-290. doi: 10.1016/j.whi.2023.12.004. Epub 2024 Feb 1. PMID 38302344
- [Result] Hoyt-Austin A, Chen MJ, Iwuagwu C, Brown SD, Fix M, Kair LR, Schwarz EB. Understanding of Lactational Amenorrhea As a Contraceptive Method Among U.S. Pregnant Women. Breastfeed Med. 2023 Aug;18(8):621-625. doi: 10.1089/bfm.2023.0105. Epub 2023 Aug 7. PMID 37578450
- [Result] Cameron NA, Begna H, Schwarz EB. Blood Pressure Monitoring and Knowledge in the First Year after a Hypertensive Disorder of Pregnancy. J Womens Health (Larchmt). 2025 Apr;34(4):485-490. doi: 10.1089/jwh.2024.0798. Epub 2024 Dec 9. PMID 39648739
- See also: Learn more or sign up for the study here! — https://studypages.com/s/healthy-moms-study-765273/